CLINICAL TRIAL: NCT05555394
Title: Effectiveness of a Rehabilitation Programme Based on Lifestyle Changes and Self-care in Patients Diagnosed With Fibromyalgia: Neuroinflammatory and Neuropsychological Biomarkers.
Brief Title: Body Awareness Therapy and Biomarkers in Fibromyalgia
Acronym: BATBF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Consorci Sanitari de l'Anoia (Other)
Responsible Party: Principal Investigator, Cristina Bravo, Postdoctoral Researcher, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04 University of Lleida
Record Dates: First submitted 2022-09-14; First posted 2022-09-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia
Keywords: Body awareness therapy; physical therapy; serotonin; cortisol
MeSH Terms: conditions — Fibromyalgia | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: clinical trial randomized allocated controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the patients don't know what intervention of study. Investigator don't know the allocation of patients outcomes assessor don't know the allocation of patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Basic Body Awareness Therapy (Experimental): the Basic Body Awareness Therapy is usual therapy of physiotherapy in mental health in nord europe. BBAT is based in twelve movements and massage that improve the movements quality of patient, also improves other movement qualities like biomechanical, physiologic, socio-cultural and existential
  Interventions: Other: Basic Body Awareness Therapy
- Stretching group (Active Comparator): Stretching exercise will be developed in control group in order to blind the intervention of interest. It will consist in analytic stretching of trunk, upper and lower limb.
  It will last around 45 min twice a week during 12 weeks.
  Interventions: Other: Stretching Exercise

INTERVENTIONS:
Other: Basic Body Awareness Therapy — The intervention will be twice a week during 12 weeks. It lasts 90 min of movements of daily life, massage and self-reflections.
  Other Names: BBAT
  Arms: Basic Body Awareness Therapy
Other: Stretching Exercise — It consists in stretching movements of whole body
  Arms: Stretching group

SUMMARY:
A randomized trial of Basic Body Awareness Therapy (BBAT) is applied in fibromyalgia patients as compared with a control intervention consisting of stretching. Sessions of BBAT lasted 90 min each and took place twice a week form 12 weeks. The primary end point is a change in the biomarkers and neurotransmitters and the Fibromyalgia Impact Questionnaire and the secondary end points include Visual Analog Scale, State Trait Anxiety inventory, Beck Depression Inventory. All assessments will be repeated at post treatment, 12 and 24 weeks and 1 year follow-up.

DETAILED DESCRIPTION:
This work is a clinical trial of randomized and controlled groups. The hypothesis of study is that BBAT applied in patients with fibromyalgia improves, more than stretching exercises, the pain, normalization biomarkers, improve in psychological state and quality life.

The study population will be selected followed the inclusion criteria of fibromyalgia, and will be selected in Consorci Sociosanitari of Anoia, the patients will be divided in 2 groups, control and treatment group. The groups will be examined at the begin, at 2 weeks, at the end of treatment and 3, 6 and 12 months follow-up.

The dependence measurements will be biomarkers serotonin, dopamine and cortisol, also Visual Analog Scale, State Trait Anxiety Inventory (STAI A/R), Beck Depression Inventory (BDI-II) and Fibromyalgia Impact Questionnaire (FIQ). The independence measurements will be demographic items: sex, age, country, level of studies, social status...

ELIGIBILITY:
Inclusion Criteria:

* whose diagnosed of fibromyalgia almost 6 months before
* whose could be in different position such as lying, sitting, and stand-up

Exclusion Criteria:

* whose are diagnosed of disease that it worse the pain
* pregnancy
* whose are diagnosed of other disease such as rheumatology, neurology, cardiac problems o another internal medical condition,malignant disease or acute infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Serotonin | through study completion, an average of 1 year
  Neurotransmitter neurologic
cortisol | during the procedure
  acute hormone relating stress

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | through study completion, an average of 1 year
  Assess of subjective pain of patient. It consists in a number between 0 to 10
Fibromyalgia Impact Questionnaire (FIQ) | through study completion, an average of 1 year
  Questionnaire about the impact of symptoms of Fibromyalgia in daily life. It measures 21 items with a total score between 0 to 100. The main average is 50.
Beck Depression Inventory- II (BDI-II) | through study completion, an average of 1 year
  Questionnaire for assess the depression of patient. It consists in 21 items with scale ranking from 0-3 with a total score from 0-63. A score between 10-18 corresponds to mild to moderate depression, further than 30 corresponds to severe depression
State Trait Anxiety Inventory (STAI) | through study completion, an average of 1 year
  Questionnaire for assess the anxiety of patient. It consists in 20 questions that score range from 20 to 80. The higher scores correlating with greater anxiety. The questionnaire provide information about state (how a person is feeling at the time) and trait (how people feel across typical situations that everyone experiences on a daily basis)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Consorci Sanitari de l'Anoia, Igualada, Barcelona
  - Cristina Bravo Navarro, Igualada, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atasever M, Namli Kalem M, Sonmez C, Seval MM, Yuce T, Sahin Aker S, Koc A, Genc H. Lower serotonin level and higher rate of fibromyalgia syndrome with advancing pregnancy. J Matern Fetal Neonatal Med. 2017 Sep;30(18):2204-2211. doi: 10.1080/14767058.2016.1243096. Epub 2016 Nov 29. PMID 27696917
- [Background] Busch AJ, Webber SC, Brachaniec M, Bidonde J, Bello-Haas VD, Danyliw AD, Overend TJ, Richards RS, Sawant A, Schachter CL. Exercise therapy for fibromyalgia. Curr Pain Headache Rep. 2011 Oct;15(5):358-67. doi: 10.1007/s11916-011-0214-2. PMID 21725900
- [Background] Bravo C, Skjaerven LH, Espart A, Guitard Sein-Echaluce L, Catalan-Matamoros D. Basic Body Awareness Therapy in patients suffering from fibromyalgia: A randomized clinical trial. Physiother Theory Pract. 2019 Oct;35(10):919-929. doi: 10.1080/09593985.2018.1467520. Epub 2018 May 3. PMID 29723080
- [Background] Bravo C, Skjaerven LH, Guitard Sein-Echaluce L, Catalan-Matamoros D. Effectiveness of movement and body awareness therapies in patients with fibromyalgia: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2019 Oct;55(5):646-657. doi: 10.23736/S1973-9087.19.05291-2. Epub 2019 May 15. PMID 31106558
- [Background] Coppieters I, Cagnie B, Nijs J, van Oosterwijck J, Danneels L, De Pauw R, Meeus M. Effects of Stress and Relaxation on Central Pain Modulation in Chronic Whiplash and Fibromyalgia Patients Compared to Healthy Controls. Pain Physician. 2016 Mar;19(3):119-30. PMID 27008285